CLINICAL TRIAL: NCT02865031
Title: Intravitreal Decorin Preventing Proliferative Vitreoretinopathy in Perforating Injuries: a Pilot Study.
Brief Title: Dacorin for Proliferative Vitreoretinopathy
Acronym: Dacorin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tamer Ahmed Macky, Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Dacorin
Record Dates: First submitted 2016-08-06; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: PVR
MeSH Terms: interventions — Decorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decorin (Experimental): Intravitreal injection of 200-400 ug of Decorin.
  Interventions: Drug: Decorin

INTERVENTIONS:
Drug: Decorin — Intravitreal Injection following ocular trauma to prevent scar tissue formation.

SUMMARY:
Purpose: To determine the safety, tolerability, and efficacy of human recombinant decorin protein, a transforming growth factor ß (TGFß) inhibitor in preventing proliferative vitreoretinopathy (PVR) in patients with perforating globe injuries.

Methods: This is a prospective, single-center, open-label, interventional case series. A single intravitreal injection of decorin 200ug (n=4) and 400ug (n=8) was given within 24 hours of injury. Pars plana vitrectomy with silicone oil injection was done if indicated. ERG was done before injections, at day 10, and 3 months. Serial plasma decorin levels were assessed before injections, day 3, 5, and 10 post-injection. Clinical assessment included globe survival, retinal attachment rate, and PVR evaluation.

DETAILED DESCRIPTION:
This is prospective, single-center, open-label, interventional case series. Twelve patients with open globe injuries presenting to the causality department at Kasr Al Ainy Teaching Hospital, Cairo University, were enrolled in our study. Those patients were assigned to Ocular Trauma Score category 1 or 2 in which the visual prognosis after treatment is poor (Category 1 prognosis: 74% no light perception, 15% light perception to hand movements, Category 2 prognosis: 27% no light perception, 26% light perception to hand movements) (31).

An informed consent was obtained from the participant prior to the conduct of any study procedure. The participant was adequately informed about the study, understood risks, benefits and alternative treatments, and voluntarily agreed to participate in the study. He / She was given ample time to consider participation and had his / her questions addressed in a satisfactory manner before agreeing to participate and signing the informed consent form. Participants were free to choose to withdraw from the study at any time without any responsibility, even if the study has not been completed.

Pre-operative Evaluation: 1. Baseline systemic examination: including clinical evaluation, complete blood picture, liver function tests and kidney function tests. 2. Full ocular examination: All patients were subjected to complete ophthalmological examination including: Best corrected visual acuity (according to the Snellen VA chart). Slit lamp examination. 3. CT scan (Sytec and BrightSpeed; GE Healthcare, Milwaukee, Wis): Unenhanced CT of the orbits was performed; axial, coronal and sagittal views with contiguous 2-mm-thick sections.

4. Full Field ERG using a full field flash Ganzfeld stimulator (Roland Consult, Electrophysiologic Diagnostic Systems, Wiesbaden, Germany): The ISCEV-ERG GF program was used to record standard ERGs. All responses were differentially amplified, displayed on an oscilloscope, digitized and stored on a compact disc. An adjustable voltage window was used to reject records contaminated by artifacts.

Dark adapted ERG responses were obtained after a minimum of 30 minutes of dark adaptation and included an isolated rod, standard flash (maximal) response, and oscillatory potentials. Light adapted responses included a single white flash and 30-Hz flicker. ERG amplitudes and implicit time values were measured according to recommendations by the International Society for Clinical Electrophysiology of Vision.

The time interval between the time of injury and the time of primary repair was recorded.

Decorin Injection:

One dose of 200 µg/0.1ml or 400 µg/0.1ml Recombinant Human Decorin (R&D Systems, Inc., Minneapolis, MN, USA) are to be evaluated in this study and is to be injected intravitreally. Those doses were reported to be effective and safe in a rabbit model of traumatic PVR. Considering the difference of the vitreous volume between human and rabbits; three times larger in the former; the dose was expected to be tolerable in human. The drug was injected within 48 hours after the trauma taking all the safety measures for intravitreal drug injections according to the The Royal College of Ophthalmologist guidelines of intravitreal injections procedure 2009.

Surgical management:

Surgery is done in two steps:

Step I: Primary repair:

Initial repair of the globe is to be done at the time of presentation. The globe is explored for injuries. The severity of the trauma is evaluated and documented to insure that the case fulfill the inclusion criteria of the study.

Step II: Secondary intervention:

Delayed vitrectomy at the tenth day after the injury was done with silicon oil temponade.

Primary repair: General anaesthesia. Sterilization with betadine 10% for the eye lids. Application of sterile drapes and wire speculum. Conjunctival dissection and removal of any tenon tissue at edges of the inlet scleral wound. Rectus muscle is hooked and cut whenever needed for proper exposure of the wound. Vitrectomy was done for any prolapsed vitreous from the wound. Scleral wound was sutured using 7/0 vicryl suture on reverse cutting needle. Conjunctiva was closed with inverted knot using 7/0 vicryl suture.

Post Primary Repair Follow Up: 1. Systemic follow up: including clinical evaluation, complete blood picture, liver function tests and kidney function tests at the tenth day. 2. Ocular examination follow up: Slit lamp examination accessing; Sutured wound. Anterior chamber cells and flare; Intraocular pressure. Follow up ERG: at tenth day. Measuring plasma Decorin level at third, fifth, eighth and tenth day. Ocular Ultrasound: to detect site of exist, presence of retinal detachment, state of posterior hyaloid, suprachoroidal hemorrhage, subretinal hemorrhage and presence of intraocular foreign body.

Pars Plana Vitrectomy: General anaesthesia. Sterilization with betadine 10% for the eye lids and betadine eye drops 5% for the surface of the globe. Application of sterile drapes and wire speculum. 23G vitrectomy system was used. Using one step technique, the 23G cannulas were inserted obliquely after minimal displacement of the intact conjunctiva using a pressure plate for globe fixation and as a measure. The infusion line was inserted into the infero-temporal cannula. Before opening the infusion, a vitreous sample was taken by vitrectomy cutter with the aspiration line plugged to a 5ml syringe to measure vitreous Decorin level. Hemorrhagic anterior hyaloid behind the posterior capsule was removed, utilizing light from operating microscope, taking care not to injure posterior capsule. Infusion cannula was verified that it was in vitreous cavity not in the suprachoriod space. Non-contact wide-angle viewing system binocular indirect ophthalmomicroscope (BIOM) was used for visualization. Hemorrhagic vitreous gel was excised, layer by layer, taking care not to injure the retina especially in cases associated with retinal detachment. The hemorrhagic tissue over the posterior exist wound was trimmed by the vitrectomy probe. The vitrectomy probe, with the vacuum mode, was used to look for adherent posterior cortical vitreous. The probe was placed just above the optic disc with the aspiration port directed away from the macular area. Vacuum was gradually increased until the cortical vitreous was engaged in the aspiration port. The probe was withdrawn anteriorly while gradually increasing the vacuum until the posterior hyaloid was detached and elevated from the posterior pole. This was assured by observing the circular wave spreading peripherally. Next, the detached posterior hyaloid engaged in the aspiration port, was peeled from posterior to anterior. The vitreoretinal interface during surgical posterior hyaloid peeling was closely observed, so that peeling was stopped once strong attachments were encountered for fear of creating retinal tear. Whenever possible, peeling was continued till the posterior border of vitreous base. To ensure complete detachment of the posterior hyaloid, triamcinolone acetinoide was injected gently into the mid vitreous cavity. Posterior cortical vitreous still adherent to the retinal became highlighted. The later was removed using vacuum generated at the probe aspiration port, soft tip back-flush flute needle or by using Tano's scrapper. If there is retinal detachment, PFCL was injected gently through a small bored blunt cannula directed towards optic disc, while lowering the intraocular pressure, to flatten the already mobilized retina over the posterior pole. Subretinal fluid was drained through existing retinal breaks or retinotomies when necessary. Vitrectomy for the vitreous base was performed meticulously 360 degrees with scleral indentation accomplished by the assistant. The IOP was lowered during base vitrectomy to reduce counter-resistance and allow easy depression of the sclera. The vitreous cutter was set at 5,000 cuts per minute and the suction was adjusted with the foot pedal. The sclera was depressed gently with the narrow shaft of the scleral depressor while the suction was increased. Both hands were used to remove the vitreous base; vitrectomy at the vitreous base from the 6- to 12-o'clock position was performed with the vitreous cutter held with the right hand, and that from the 12- to 6-o'clock position was performed with the left hand. Endolaser photocoagulation was applied around posterior exist site, 360 degrees and to all retinal breaks. Silicone oil was injected through the infusion cannula. Closure of two sclerotomies. Removal of the infusion cannula and closure of the third sclerotomy. Eye patching. Adjuvant scleral buckling was not performed in any case. Patients were instructed to maintain the appropriate position for 1 week following surgery.

Post-operative follow-up: Full ophthalmological examination was done on the first day post-operatively then at 1st week and 1st month. Examination included: Best corrected visual acuity (according to the Snellen VA chart). Slit lamp examination. Assessment of IOP. Dilated fundus examination with binocular indirect slit-lamp biomicroscopy using (Super Field lens; VOLK, Mentor, Ohio, USA).After 3 months, silicone oil was removed. The retinal status was evaluated again, after silicone removal, with binocular indirect slit-lamp biomicroscopy using (Super Field lens; VOLK, Mentor, Ohio, USA). Furthur assessment of the retina was done, functionally by ERG and anatomically by sweept source OCT. SS-OCT (DRI OCT-1, Topcon, Japan) using radial and raster scans was done over the macula and the edge of the posterior exist scar (Figure 31). The investigators evaluated the presence or absence of any epi or sub retinal membranes, vitreoretinal interface abnormalities, intra-retinal fluid, subretinal fluid, the status of the IS/OS junction and ELM.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years old
* Perforating Ocular Injuries zone 2 and 3.
* ERG of the affected eye was at least 50% of the unaffected fellow eye.

Exclusion Criteria:

* No concomitant ocular disease.
* No pervious ocular surgery.
* No systemic organ failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Electrophysiological tests ERG a and b implicit time and latency | 3 months

SECONDARY OUTCOMES:
Scar tissue formation graded 0-4 grades | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdullatif AM, Macky TA, Abdullatif MM, Nassar K, Grisanti S, Mortada HA, Soliman MM. Intravitreal decorin preventing proliferative vitreoretinopathy in perforating injuries: a pilot study. Graefes Arch Clin Exp Ophthalmol. 2018 Dec;256(12):2473-2481. doi: 10.1007/s00417-018-4105-7. Epub 2018 Aug 20. PMID 30128605